CLINICAL TRIAL: NCT04175379
Title: The Effect of Permissive Hypercapnia on Oxygenation and Post-operative Pulmonary Complication During One-lung Ventilation : Prospective, Randomized Controlled Study
Brief Title: The Effect of Permissive Hypercapnia on Oxygenation and Post-operative Pulmonary Complication During One-lung Ventilation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 4-2019-0904
Record Dates: First submitted 2019-11-15; First posted 2019-11-25 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Thoracic Surgery

STUDY DESIGN:
Intervention Model Description: Random sampling using random numbers is divided into three groups, and the ratio of each group is 1: 1: 1.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Patients, care givers and outcomes assessors are blinded. The investigator should not be included in the blind because they need to adjust the ventilator settings.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- group 40 (Experimental): In group 40, target PaCO2 is 40 during surgery
  Interventions: Other: group 40
- group 50 (Experimental): In group 50, target PaCO2 is 50 during surgery
  Interventions: Other: group 50
- group 60 (Experimental): In group 60, target PaCO2 is 60 during surgery
  Interventions: Other: group 60

INTERVENTIONS:
Other: group 40 — During surgery, the TV(tidal volume) should maintain 6ml/kg (ideal body weight). After position change and OLV(one lung ventilation) for operation, each patient adjusts RR(respiratory rate) to reach target PaCO2 40 ± 5mmHg. Hemodynamic records and arterial blood tests are performed at the following times: After tracheal intubation, 15 minutes after in two lung ventilatory state at the supine position (T0), after 30 minutes reaching to the target PaCO2 by adjusting RR at the lateral position starting one lung ventilation (T1), and after 60 minutes while maintaining target PaCO2 (T2).
  Arms: group 40
Other: group 50 — During surgery, the TV(tidal volume) should maintain 6ml/kg (ideal body weight). After position change and OLV(one lung ventilation) for operation, each patient adjusts RR(respiratory rate) to reach target PaCO2 50 ± 5mmHg. Hemodynamic records and arterial blood tests are performed at the following times: After tracheal intubation, 15 minutes after in two lung ventilatory state at the supine position (T0), after 30 minutes reaching to the target PaCO2 by adjusting RR at the lateral position starting one lung ventilation (T1), and after 60 minutes while maintaining target PaCO2 (T2).
  Arms: group 50
Other: group 60 — During surgery, the TV(tidal volume) should maintain 6ml/kg (ideal body weight). After position change and OLV(one lung ventilation) for operation, each patient adjusts RR(respiratory rate) to reach target PaCO2 60 ± 5mmHg. Hemodynamic records and arterial blood tests are performed at the following times: After tracheal intubation, 15 minutes after in two lung ventilatory state at the supine position (T0), after 30 minutes reaching to the target PaCO2 by adjusting RR at the lateral position starting one lung ventilation (T1), and after 60 minutes while maintaining target PaCO2 (T2).
  Arms: group 60

SUMMARY:
Permissive hypercapnia increased the survival rate in patients with acute respiratory distress syndrome (ARDS) who required mechanical ventilation in critical care medicine. This has been explained by its association with ventilator induced lung injury. Since then, a protective lung ventilation strategy has been very important, with a low tidal volume of 4-6 ml/kg. Patients undergoing surgery will inevitably require mechanical ventilation. In particular, patients undergoing one lung ventilation for thoracic surgery may have increased airway pressure and a greater chance of ventilator induced lung injury. Recently, protective lung ventilation has been applied to patients undergoing one ung ventilation during thoracic surgery. The purpose of this study is to evaluate the difference in the degree of pulmonary oxygenation and the incidence of postoperative pulmonary complications in hypercapnia induced by controlling the respiratory rate with a constant tidal volume.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients aged 40-80 years who are planning to have thoracoscopic single lobectomy or segmentectomy with one lung ventilation during surgery.
2. American Society of Anesthesiologists (ASA) classification 1~3

Exclusion Criteria:

1. patients with heart failure (NYHA class III~IV)
2. patients who are having moderate obstructive lung disease or restrictive lung disease
3. Low DLCO (< 75%)
4. patients with brain disease history or increased ICP
5. patients with pulmonary hypertension (mean PAP>25mmHg)
6. patients with liver disease (AST level ≥100 IU/mL or ALT ≥ level 50 IU/L) or kidney disease (Creatine level ≥ 1.5 mg/dL)
7. patients with pre-existing hypercapnia or metabolic acidosis
8. body mass index (BMI) > 30 kg/m2
9. patients who have had contralateral lung surgery
10. patients who cannot read explanation and consent form
11. patients who are pregnant

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 279 (Estimated)
Dates: Start 2019-11-25 (Actual); Primary Completion 2021-08 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
PaO2/FiO2 ratio | about 60 minutes after reaching to the target PaCO2 (T2)
  (arterial oxygen partial pressure / fractional inspired oxygen) at the time of T2 (PaO2 of ABGA/FiO2) T2

SECONDARY OUTCOMES:
Post-op complication: desaturation event | first 3 days after surgery
  desaturation event (<90%) the first 3 days after surgery
Post-op complication: oxygen therapy | first 2~7 days after surgery
  necessity of oxygen therapy within the first 2~7 days after surgery hospitalized days, ICU days, expire
Post-op complication | 30 days after surgery
  The presence or absence of post operative complication like pneumonia, acute lung injury, re-intubation, ICU admission, ventilator care, empyema, broncho-pleura fistula, air-leakage, pleural effusion, pulmonary embolism, tracheostomy, wound infection, AKI, MI, etc.
Post-op complication: hospitalized days | 30 days after surgery
  length of hospitalized stays CU days, expire
Post-op complication: ICU days | 30 days after surgery
  length of ICU stays
Dead | 30 days after surgery
  patient has been dead or not

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anaesthesiology and Pain Medicine, Anaesthesia and Pain Research Institute, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Joe YE, Lee CY, Kim N, Lee K, Kang SJ, Oh YJ. Effect of permissive hypercarbia on lung oxygenation during one-lung ventilation and postoperative pulmonary complications in patients undergoing thoracic surgery: A prospective randomised controlled trial. Eur J Anaesthesiol. 2023 Sep 1;40(9):691-698. doi: 10.1097/EJA.0000000000001873. Epub 2023 Jul 15. PMID 37455644